CLINICAL TRIAL: NCT06093958
Title: Paradoxical Response to Chest Wall Loading in Mechanically Ventilated Patients: Incidence, Mechanism, and Novel Techniques for Detecting it at the Bedside
Brief Title: Paradoxical Response to Chest Wall Loading in Mechanically Ventilated Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively closed by IRB after continuing review was never submitted and no patients enrolled.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A21-280
Record Dates: First submitted 2021-11-08; First posted 2023-10-23 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2021-11

CONDITIONS: ARDS; COVID-19; Mechanical Ventilation Pressure High; Ventilator-Induced Lung Injury
MeSH Terms: conditions — COVID-19; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Chest wall loading (Experimental): All patients who are receiving mechanical ventilation and are passive on the ventilator will have chest wall loading performed to identify whether there is a paradoxical decrease in lung compliance.
  Interventions: Diagnostic Test: Manual loading of the chest wall

INTERVENTIONS:
Diagnostic Test: Manual loading of the chest wall — The chest wall will be loaded by either compression of the abdominal wall, compression of the lumbar spine, or compression of the sternum.

SUMMARY:
The purposes of our study are to: 1) determine the incidence of paradoxical response to chest wall loading in mechanically ventilated patients; 2) identify sub-populations in which it is most likely to occur (e.g., severe ARDS); and 3) standard the bedside procedure for demonstrating this physiology.

DETAILED DESCRIPTION:
Mechanical ventilation can be a life-saving intervention for patients with respiratory failure, but the acutely injured lung is vulnerable to further damage if positive pressure ventilation is not employed judiciously. "Lung protective ventilation" encompasses a group of practices intended to minimize ventilator-induced lung injury (VILI) and includes the delivery of low tidal volumes (to minimize dynamic lung strain) and the prevention of injuriously high airway pressures (to minimize lung stress). The prone position, which compresses (or "loads") the chest wall, more evenly distributes volume and pressure, mitigates the damaging effects of stress/strain, and improves clinical outcomes in patients with severe respiratory failure from adult respiratory distress syndrome (ARDS).

Chest wall loading would not be expected to produce these beneficial effects in the supine position-quite the opposite; it usually results in net volume loss and higher airway pressures in response to an unchanging tidal volume. A paradoxical response to chest wall loading, leading to decreased airway pressures, however, was recently reported in a group of patients with advanced lung disease secondary to COVID-19. In this cohort, a paradoxical decrease in airway pressures was elicited during a brief period of manual compression of the abdomen.

This maneuver, which is non-invasive, free of cost, and gives real-time information, may have important diagnostic (and potentially therapeutic) implications for ventilator management in patients with respiratory failure.

ELIGIBILITY:
Inclusion Criteria: Non-surgical patients admitted to the ICU at Regions Hospital (St. Paul, MN) or Methodist Hospital (St. Louis Park, MN), receiving mechanical ventilation for any reason, and breathe passively during mechanical ventilation

Exclusion Criteria:

1. Age < 18 years old
2. Pregnancy at the time of their inclusionary hospitalization
3. Recent (< 30 days) abdominal or chest wall surgery (including spine)
4. Recent (< 30 days) abdominal or chest wall trauma (including spine)
5. Traumatic brain injury, intracranial bleed, or recent neurologic surgery
6. Family member or representative not available to provide informed consent
7. Not passive while receiving mechanical ventilation support
8. Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Lung compliance (mL/mmHg) | 20 minutes total in measure duration.
  Does lung compliance improve (ie, increase) with an intervention (chest wall loading) that decreases chest wall compliance/reduces lung volume.

CONTACTS AND LOCATIONS:
Overall Officials: John Selickman, MD, Principal Investigator — University of Minnesota
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
This study did not enroll any participants so there is no IPD to be shared.